CLINICAL TRIAL: NCT02876822
Title: Safety and Efficacy of Single, High Dose Vitamin D Replacement in Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: High Dose Vitamin D Replacement in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Step 1 enrollment complete.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2193
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Experimental): Enrolled subjects will receive one observed oral vitamin D dose (based on current vitamin D status and rounded to the nearest 5000IU) within 2 weeks prior to their HSCT.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Other Names: cholecalciferol

SUMMARY:
The purpose of this study is to test the efficacy and safety of high dose vitamin D therapy among HSCT patients in a tiered, step-wise manner (step one/two) in order to define treatment doses capable of providing vitamin D sufficiency.

DETAILED DESCRIPTION:
Vitamin D deficiency is common in childhood and has been associated with increased incidence of graft versus host disease (GVHD) and decreased survival in patients undergoing hematopoietic stem cell transplantation (HSCT). Recently, quality improvement efforts to correct serum vitamin D levels among inpatients at CCHMC who have already received HSCT and who were vitamin D deficient suggest that current recommended doses of vitamin D are inadequate to treat vitamin D deficiency. Possible hindrances to vitamin D treatment in the HSCT population include malabsorption related to gut GVHD, mucositis, increased requirement for calcium and/or vitamin D, kidney disease, liver disease, and infection. Single, high dose vitamin D treatment (stoss-therapy) has been utilized effectively to treat rickets and other chronic illnesses such as cystic fibrosis in children. The investigators hypothesize that stoss-therapy provided orally prior to transplantation will result in rapid and sustained correction of vitamin D deficiency in children who require HSCT. The investigators propose to test the efficacy and safety of high dose vitamin D therapy among HSCT patients in a tiered, step-wise manner (step one/two) in order to define treatment doses capable of providing vitamin D sufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Step 1: Patients who are preparing for HSCT, 25OHD level (<50 ng/mL), and no prior history of HSCT.
* Step 2: Patients who are preparing for HSCT 25OHD level (<50 ng/mL).

Exclusion Criteria (both Step 1 and Step 2):

* Patients with history of pathologic fractures,
* uncorrected hypocalcemia or hypophosphatemia,
* known history of nephrocalcinosis or nephrolithiasis,
* current granulomatous disease,
* those currently in ICU.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Serum 25OHD level | Weekly for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howell, MD, Principal Investigator — Cincinnati Children's Hosptial Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No